CLINICAL TRIAL: NCT00094393
Title: Clinical Investigations Into Hutchison-Gilford Progeria Syndrome
Brief Title: Clinical Studies of Progeria
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050004; 05-HG-0004
Record Dates: First submitted 2004-10-16; First posted 2004-10-18 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2018-05-22

CONDITIONS: Progeria
Keywords: Ageing; Atherosclerosis; Lamin A; Lipodystrophy; Growth Impairment; Premature Aging; Hutchinson-Gilford Progeria Syndrome; HGPS
MeSH Terms: conditions — Progeria; Atherosclerosis; Autosomal Emery-Dreifuss Muscular Dystrophy; Lipodystrophy; Aging, Premature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
This study will examine children with Hutchinson-Gilford Progeria syndrome, a genetic disease that causes many changes to the body over time, including heart disease, bone changes, hair loss, and joint and skin changes. Often called a "premature aging" disease, progeria does not mimic aging completely. This study will examine which body systems are affected in progeria and how each system is affected over time in order to try to develop new treatments.

Patients with progeria who are between 6 months and 70 years of age and who are able to travel to the NIH in Bethesda, Md., may be eligible for this 5- to 10-year study.

Participants come to the NIH Clinical Center for evaluation every 2 years. Each 4-5 day visit includes the following tests and procedures:

* Medical history and physical examination
* Blood tests to analyze cardiovascular risk factors, blood counts, blood chemistries, and for research
* Urine tests for sugar and proteins
* Photographs to study growth problems
* X-ray studies to determine bone density and body composition, such as body fat and muscle
* Electrocardiogram (EKG) and echocardiogram (heart ultrasound) to study the heart and blood vessels
* Lung function tests to measure energy consumption and lung capacity
* Skin biopsy (surgical removal of a small skin sample) to examine cellular changes
* Hearing tests
* Eye examination to evaluate eyesight, eye pressure and structures of the eye
* Physical therapy evaluation with stretching and exercises to measure how the joints bend and straighten
* Dental examination, including X-rays
* Meeting with a nutritionist who will track the patient's food intake and take body measurements
* Magnetic resonance imaging (MRI) for patients who are old enough to undergo the procedure without sedation. This test uses a magnetic field and radio waves to examine body organs. For this test, the patient must lie still in the scanner, a narrow cylindrical tube.

Patients are provided the results of their medical tests. Information about the patient is submitted to the PRF Cell and Tissue Bank in Peabody, Massachusetts.

DETAILED DESCRIPTION:
Hutchison-Gilford Progeria Syndrome (HGPS) is a rare "premature aging" disease in which children die of severe atherosclerosis at an average age of thirteen years (range 8-20 years). Children with HGPS appear healthy at birth, but within months display signs of growth failure, lipodystrophy, hair loss, and aged skin. Within just a few years they exhibit boney abnormalities including osteoporosis and resorption, coax valga and hip dislocation. The final height approximates 3 feet. Mortality is caused by generalized artherosclerosis leading to strokes and heart attacks. The gene defect causing HGPS has recently been identified as a single base mutation in the gene LMNA, coding for the nuclear protein Lamin A. The spectrum of effects of this gene defect on cellular function, and how these effects culminate in the HGPS disease phenotype, remain to be elucidated. Furthermore, no in-patient multisubject clinical evaluation of children with HGPS has ever been performed, and no therapy exists for any of the complications of HGPS. Hence, baseline studies are critical to determine the extent of organ involvement in HGPS, evaluate disease progression, and design clinical trials of potential treatments. The purpose of this study is to longitudinally investigate the disease characteristics of HGPS using state-of the-art measures of cardiovascular function, comprehensive laboratory testing, in vitro cell culture studies, and extensive medical consultations. HGPS patients will be admitted to the NIH Clinical center as inpatients for approximately 5 days every two years. The information emanating from the proposed studies will assist in assuring appropriate care for children with HGPS, provide a better understanding of the variations in phenotype of HGPS, and stimulate new research into HGPS and the aging diseases associated with HGPS, such as atherosclerosis. These studies will also allow us to evaluate new clinical outcome parameters and to design appropriate therapeutic interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Inclusion criteria consist of male and female children of all ethnic groups with the diagnosis of HGPS.
* An individual in whom a clinical diagnosis of HGPS has been

verified by Dr. Gordon will be eligible for this protocol.

EXCLUSION CRITERIA:

- Exclusion criteria consist of patients below 6 months and over 70 years of age. Another exclusion is the inability to travel to the NIH due to advanced cardiovascular disease, as reflected by unstable angina, congestive heart failure, or other serious symptoms.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-10-14; Study Completion 2018-05-22

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] DeBusk FL. The Hutchinson-Gilford progeria syndrome. Report of 4 cases and review of the literature. J Pediatr. 1972 Apr;80(4):697-724. doi: 10.1016/s0022-3476(72)80229-4. No abstract available. PMID 4552697
- [Background] Pesce K, Rothe MJ. The premature aging syndromes. Clin Dermatol. 1996 Mar-Apr;14(2):161-70. doi: 10.1016/0738-081x(95)00151-5. No abstract available. PMID 9117983
- [Background] Badame AJ. Progeria. Arch Dermatol. 1989 Apr;125(4):540-4. PMID 2649013
- [Derived] Merideth MA, Gordon LB, Clauss S, Sachdev V, Smith AC, Perry MB, Brewer CC, Zalewski C, Kim HJ, Solomon B, Brooks BP, Gerber LH, Turner ML, Domingo DL, Hart TC, Graf J, Reynolds JC, Gropman A, Yanovski JA, Gerhard-Herman M, Collins FS, Nabel EG, Cannon RO 3rd, Gahl WA, Introne WJ. Phenotype and course of Hutchinson-Gilford progeria syndrome. N Engl J Med. 2008 Feb 7;358(6):592-604. doi: 10.1056/NEJMoa0706898. PMID 18256394